CLINICAL TRIAL: NCT04725591
Title: An Open-label, Multicenter, Randomized, Crossover Study, to Assess 4 Weeks Outpatient, the Clinical Efficacy of the Diabeloop Closed-loop Glucose Control Without the Declaration of Meals Compared with the Diabeloop Closed-loop Glucose Control with the Declaration of Meals, in Adolescent Patients with Type 1 Diabetes Poorly Controlled.
Brief Title: Diabeloop for Teens
Acronym: DBL4T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A02132-37
Record Dates: First submitted 2021-01-13; First posted 2021-01-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Closed Loop; Diabetes Mellitus, Type 1; Adolescents (12 to 17 Years Old)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabeloop closed-loop glucose control session with the declaration of meals (Active Comparator): Diabeloop software (an MPC-based glucose control algorithm) running on handset associated with the six-generation glucose sensor (Dexcom G6) and MEDISAFE WITH insulin pump.
  Subjects are asked to declare their meals for 4 weeks.
  A remote monitoring system is provided in closed-loop session.
  Interventions: Device: Dexcom G6 Continuous Glucose Monitoring; Device: MEDISAFE WITH External Insulin Pump; Device: Diabeloop Software (Model predictive control); Other: Declaration of meals; Other: Remote monitoring (Telemedicine)
- Diabeloop closed-loop glucose control session without the declaration of meals (Experimental): Diabeloop software (an MPC-based glucose control algorithm) running on handset associated with the six-generation glucose sensor (Dexcom G6) and MEDISAFE WITH insulin pump.
  Subjects are asked to not declare their meals for 4 weeks.
  A remote monitoring system is provided in closed-loop session.
  Interventions: Device: Dexcom G6 Continuous Glucose Monitoring; Device: MEDISAFE WITH External Insulin Pump; Device: Diabeloop Software (Model predictive control); Other: No declaration of meals; Other: Remote monitoring (Telemedicine)

INTERVENTIONS:
Device: Dexcom G6 Continuous Glucose Monitoring — Collection of glucose data
Device: MEDISAFE WITH External Insulin Pump — Insulin delivery
Device: Diabeloop Software (Model predictive control) — Diabeloop software embeds a regulation algorithm to automatically regulate the patient's glycaemia. It takes as input glycaemia value received every 5 minutes from the CGM and patient inputs related to meals and physical activities and it calculates the amount of insulin to be delivered. It sends this information to the pump that automatically delivers this quantity.
Other: Declaration of meals — Patient inputs related to meals
  Arms: Diabeloop closed-loop glucose control session with the declaration of meals
Other: No declaration of meals — No patient inputs related to meals
  Arms: Diabeloop closed-loop glucose control session without the declaration of meals
Other: Remote monitoring (Telemedicine) — Remote follow up by care health providers team

SUMMARY:
An open-label, three-centers, controlled, randomized, and crossover study containing 14 days of baseline period with standard of care (SOC) therapy followed by two-sessions of 4-weeks home study phase with Diabeloop closed-loop (CL) system comparing the declaration of meals and the non-declaration of meals.

ELIGIBILITY:
Inclusion Criteria:

Device-related inclusion criteria

* age 12 - <18 years (i.e 17 years and 364 days) at time of screening
* Type 1 diabetes Study-specific inclusion criteria
* Subject has a clinical diagnosis of type 1 diabetes for at least 1 year as determined via medical records or source documentation by an individual qualiﬁed to make a medical diagnosis or confirmed C peptide negative.
* An insulin pump user, or patient under Multiple Daily Injection (MDI), with or without CGM experience.
* Subject having a Glycosylated hemoglobin (HbA1c) blood value > 8 % at time of screening visit-based on analysis from local laboratory within 3 months.
* Living in an area covered by a GSM (Global System for Mobile Communications) network
* Patient not isolated, does not live alone, or has a person living nearby who has a telephone and a key to his or her home
* Patient willing to wear the system continuously throughout the study
* Must be able to speak and be literate in French, in Dutch or in German
* Having provided written assent & parents/guardian having provided written informed consent

Exclusion Criteria:

Device-related exclusion criteria

* Patient receiving a total daily dose of insulin lower than 8 U
* Patient having severe uncorrected problems of hearing and/or visual acuity
* Patient unable to understand and perform all of the instructions provided by Diabeloop SA Study-specific exclusion criteria
* Subject is unable to tolerate tape adhesive around the sensor or pump placements
* Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection)
* Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
* Is being treated for hyperthyroidism at time of screening
* Has diagnosis of adrenal insufficiency
* Has taken any oral, injectable, or intravenous (IV) steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the study
* Females who are sexually active and able to conceive will be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study as determined by investigator.
* Actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks
* Currently abusing illicit drugs
* Currently abusing marijuana
* Currently abusing prescription drugs
* Currently abusing alcohol
* Subject is using pramlintide (Symlin), DDP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of screening
* Subject has elective surgery planned that requires general anesthesia during the study
* Has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
* Plans to receive red blood cell transfusion or erythropoietin over study participation
* Diagnosed with current eating disorder such as anorexia or bulimia
* Diagnosed with chronic kidney disease that results in chronic anemia
* Hematocrit that is below the normal reference range of lab used
* Patient who has had a pancreatectomy or who has pancreatic malfunctions
* Patient with pancreatic islet transplantation or pancreas transplantation
* Patient on dialysis
* Patient with impaired hepatic functions
* Serum creatinine > 176 µmol/L
* Any other physical or psychological disease, or medication likely to interfere with the conduct of the study and interpretation of the study results as judged by the investigator.
* Pregnancy or breastfeeding
* Untreated coeliac disease (2 x ULN local laboratory)
* Untreated or unstable thyroid disease
* Subject has a history of 2 or more episodes of severe hypoglycemia, which resulted in any of the following during the 6 months prior to screening:

  * Medical assistance (i.e. Paramedics, Emergency Room or Hospitalization)
  * Coma
  * Seizures
* Subject having severe diabetic ketoacidosis in the 6 months prior to screening visit
* Impaired awareness of hypoglycemia (Gold Score > 4)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-05-19 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the time spent of the glucose level in the widened target range 3.9-10.0 mmol/L over the 2 last weeks of each cross-over period, as recorded by continuous subcutaneous glucose monitoring (CGM). | 2 weeks
  Measurement of glucose by CGM

SECONDARY OUTCOMES:
Incidence of severe hypoglycemia as defined by the ISPAD guidelines: | 10 weeks
  * Number of severe hypoglycemic episodes needing a third-party intervention
  * Number of severe hypoglycemic episodes with loss of consciousness
  * Number of hospitalizations because of a severe hypoglycemia episode
  * Number of hypoglycemic episodes, defined by any crossing of the threshold of 3.33 mmol/L, 3.9 mmol/L, 3.0mmol/L and < 2.8 mmol/L measured continuous glucose monitoring.
• Number of severe hyperglycemia episodes with beginning and end episode as measured by the Dexcom G6 CGM | 10 weeks
  o >19.4 mmol/L or significant ketosis (plasmatic ketones > 3 mmol/L) as defined by the ADA.
• Incidence of severe hyperglycemia | 10 weeks
  o Number of events requiring an emergency room visit or hospitalizations because of ketoacidosis (i.e. incidence of DKA)
• Percent of CGM time with glucose < 3.9 mmol/L | 10 weeks
  Measurement of glucose by CGM
• Percent of CGM time in glucose range 3.9-10.0 mmol/L | 10 weeks
  Measurement of glucose by CGM
• Mean CGM glucose | 10 weeks
  Measurement of glucose by CGM
• Percentage of sensor time in glucose level measured by the Dexcom G6 CGM, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am | 24 hours
  * < 2.8 mmol/L
  * < 3.0 mmol/L
  * < 3.3 mmol/L
  * < 3.9 mmol/L
• Number of hypoglycemic episodes with beginning and end of episode as measured by the Dexcom G6 CGM for at least 15 minutes | 10 weeks
  * < 3.9 mmol/L
  * < 3.0 mmol/L
  * ≤ 2.8 mmol/L
• Percentage of sensor time in glucose level measured by the Dexcom G6 CGM, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am | 24 hours
  * > 10.0 mmol/L
  * > 13.9 mmol/L
  * > 16.7 mmol/L
  * > 19.4 mmol/L
• Number of severe hyperglycemia episodes with beginning and end of episode as measured by the Dexcom G6 CGM | 10 weeks
  o > 19.4 mmol/L
• Number of serious adverse events, serious adverse device events, unanticipated adverse device effects | 10 weeks
• Risk of hypoglycemia and hyperglycemia (LBGI/HBGI) | 10 weeks
  Measurement of glucose by CGM
• Percentage of time spent in the 3.9-10.0 mmol/L target range, for the last 2 weeks of each cross-over session during nights, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am | 2 weeks
  Measurement of glucose by CGM
• Percentage of sensor time in glucose range 2.8 - 3.9 mmol/L, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am | 24 hours
  Measurement of glucose by CGM
• Percentage of sensor time in glucose range 3.9 - 7.8 mmol/L, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am | 24 hours
  Measurement of glucose by CGM
• Percentage of sensor time in glucose range 3.9 - 10.0 mmol/L, for 24 hours (12:00am-12:00am) and during the following periods: from 12:00am to 6:00am, from 6:00am to 12:00am | 24 hours
  Measurement of glucose by CGM
• Evolution of HbA1c calculated from CGM data | 10 weeks
  Measurement of glucose by CGM
• Average CGM glucose level during the entire period | 10 weeks
  Measurement of glucose by CGM
• Average fasting CGM glucose level at 6:00 am | 10 weeks
  Measurement of glucose by CGM
• Variability of the CGM glucose level | 10 weeks
  * the glycemic variation coefficient (CV) intra patient: CV < 36% CV ≥ 36%
  * Standard deviation (SD)
• Average dose of insulin used & its daily evolution during the entire study duration | 10 weeks
• Number of technical incidents leading to the interruption of the closed loop | 8 weeks
• Evolution over time of the DBL system's performance on a day-to-day and determination of the optimization delay of glycemic control | 8 weeks
  Measurement of glucose by CGM
• Evolution of the weekly average number of CHO intake (for patient with closed-loop) | 8 weeks
• Percentage of time spent in closed loop mode (i.e. DBL System with loop mode operating) | 8 weeks
• Percentage of time spent in operating mode for the Dexcom G6 CGM | 10 weeks
• Scoring of a questionnaire to evaluate the acceptance | 10 weeks
  o Diabetes Treatment Satisfaction Questionnaire (DTSQ) is a 12-item measure that enables self-reporting of the satisfaction about their current treatment. Scale is from 6 (very satisfied) to 0 (very dissatisfied).
• Scoring of a questionnaire to evaluate the acceptance | 10 weeks
  o Diabetes Technology Questionnaire (DTQ) aims to evaluate the impact of the closed-loop system use and diabetes specific quality of life measures in the study participants and their families, as well as satisfaction of system, as compared to conventional treatment options. The subject will answer by choosing from 5 suggestions : Strongly agree - Agree - Neither agree nor disagree - Disagree - Strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Beltrand, Principal Investigator — Necker Hospital
Locations (3):
- University Hospitals Leuven, Leuven, Belgium
- Necker Hospital, Paris, France
- Diabetes Center for Children and Adolescents Auf Der Bult, Hanover, Germany